CLINICAL TRIAL: NCT04854980
Title: Serologic Response to the SARS-CoV-2 MRNA-1273 Vaccine in Select Subsets of Oncology Patients - a Pilot Study
Brief Title: Serologic Response to the SARS-CoV-2 (COVID-19) MRNA-1273 Vaccine in Select Subsets of Oncology Patients
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Deepak Sahasrabudhe, Professor - Department of Medicine , Hematology/Oncology (SMD), University of Rochester
Other Study IDs: UMLT21037
Record Dates: First submitted 2021-04-20; First posted 2021-04-22 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2023-09

CONDITIONS: Covid19; Cancer
Keywords: Covid19; Cancer
MeSH Terms: conditions — COVID-19; Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Experimental:: Blood Sample Taken
  Interventions: Other: Blood Sample

INTERVENTIONS:
Other: Blood Sample — Blood sample, 2- to 5 tea spoon full (between 10 to 25 mL approximately) between 43 to 96 days after first dose of the vaccine.

SUMMARY:
To explore the immune response to the COVID-19 vaccine in cancer patients and compare to the general population.

DETAILED DESCRIPTION:
The purpose of this study is to measure the immune response to the COVID-19 vaccine in cancer patients and compare to the general population. This information can help optimize the timing of the mRNA-1273 vaccine relative to starting treatment for cancer, adding booster immunizations or incorporation of medications that to enhance the immune response.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are between 50 and 75 years of age;
* Have not had known or suspected infection with SARS-CoV-2 at any time;
* Subjects must fall into one of the following subsets of cancer patients:

  * Localized prostate cancer on radiotherapy or have completed radiotherapy in the last three months
  * Prostate cancer on androgen-deprivation therapy for biochemical recurrence
  * Colon cancer on adjuvant chemotherapy for stage III disease
  * CLL on a BTK inhibitor as a first-line single agent for at least 3 months
  * Melanoma patients on adjuvant immunotherapy with PD-1 checkpoint inhibitors for at least 3 months
* Have received both doses of SARS-CoV-2 mRNA-1273 vaccine with proof of vaccination or are scheduled to do so;
* Have at least a one-year life expectancy;
* Prior radiation therapy is allowed, as long as it was completed more than 6 months prior to vaccination

Exclusion Criteria:

* Subjects have a known hypersensitivity to a vaccine component;
* Have had known or suspected infection with SARS-CoV-2 at any time;
* Are organ transplant recipient on immunosuppression;
* Had received or are scheduled to receive a live virus vaccine in the period from 4 weeks prior to Dose 1 through 28 days post second dose;
* Had received or are scheduled to receive an inactivated vaccine in the period ranging from 7 days prior to Dose 1 through 7 days post second dose;
* Received high-dose corticosteroids at any time after receiving the vaccine;
* Are unable to give informed consent;
* Are receiving treatment for CLL with another agent (such as rituximab) in addition to a BTK inhibitor

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects are between 50 and 75 years of age
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
Immunological response to the vaccine | 1 year
  Vaccine response, as determined by blood concentrations of serum IgG reactive to the RBD domain of spike protein from the original SARS-CoV-2 virus will be measured by ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States